CLINICAL TRIAL: NCT05939245
Title: Comparison of Plasma Neutrophil Gelatinase-Associated Lipocalin (pNGAL) Level in De-Resuscitation With Furosemide Group and Control Group as a Predictor of Sepsis in Acute Kidney Injury Patients in the ICU Within 48 Hours of Treatment
Brief Title: Comparison of Plasma Neutrophil Gelatinase-Associated Lipocalin (pNGAL) Level in De-resuscitation With Furosemide Group and Control Group
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dita Aditianingsih, Principal investigator, Anesthesiologist Consultant, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IndonesiaUAnes042
Record Dates: First submitted 2023-06-25; First posted 2023-07-11 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Acute Kidney Injury Due to Sepsis
Keywords: De-resuscitation; Furosemide; pNGAL; SAKI
MeSH Terms: interventions — Furosemide

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Administration of continuous furosemide intravenous (Experimental)
  Interventions: Procedure: Furosemide Injection
- Administration of continuous placebo intravenous (Placebo Comparator)
  Interventions: Procedure: Placebo Injection

INTERVENTIONS:
Procedure: Furosemide Injection — Continuous infusion of furosemide is administered starting at 2 mg/hour and can be titrated until the target urine output of 1-2 cc/kg/hour is achieved for 48 hours. In case of hypotension (MAP <65 mmHg), norepinephrine is administered with titration starting at a dose of 0.05 mcg/kg/minute, along with a fluid loading of 4 cc/kg body weight or 300 cc within 5-10 minutes, until the target MAP of ≥65 mmHg is reached for 48 hours.
  Arms: Administration of continuous furosemide intravenous
Procedure: Placebo Injection — Continuous infusion of placebo fluid is administered at a rate of 2 mL/hour. In case of hypotension (MAP <65 mmHg), norepinephrine is administered with titration starting at a dose of 0.05 mcg/kg/minute, along with a fluid loading of 4 cc/kg body weight or 300 cc within 5-10 minutes, until the target MAP of ≥65 mmHg is reached for 48 hours.
  Arms: Administration of continuous placebo intravenous

SUMMARY:
The impact of early de-resuscitation with furosemide on patients with sepsis-related acute kidney injury using pNGAL as the parameter of acute kidney injury.

DETAILED DESCRIPTION:
Sepsis-related acute kidney injury (SAKI) is a complication leading to morbidity and mortality in septic patients. Some 50% of AKI patients in the Intensive Care Unit (ICU) are sepsis patients, which is the highest cause of death in the ICU. In sepsis, there is systemic inflammation that causes endothelial damage, which manifests in capillary leakage. Fluid accumulation that has occurred since the patient came to the hospital due to a capillary leak in sepsis and is exacerbated by fluid resuscitation has a negative impact on the kidneys. Therefore, the aim of this study was to assess the effectiveness of early de-resuscitation using furosemide on the incidence of AKI in septic patients using pNGAL as a parameter of AKI.

This study used a double-blind, randomized clinical trial design. This study was conducted on septic patients with a cumulative balance of >1500 mL/day and urine output of 0.8 cc/kg/hour in the ICU of Dr. Cipto Mangunkusumo National Central Public Hospital in the July-December 2023 period. pNGAL levels were checked at the 0th and 48th hours of ICU care. A total of 48 subjects were divided into 2 groups: 24 patients in the treatment group were given a continuous injection of furosemide at 2 mg/hour, and 24 patients in the control group were given a placebo injection at 2 mg/hour. The patient's condition will be followed after the ICU stay for up to 28 days to record the need for renal replacement therapy and death.

ELIGIBILITY:
Inclusion Criteria:

* Sepsis patients with a cumulative balance of >1500 mL/day and urine output <0.8 cc/kg/hour.

Exclusion Criteria:

* Has undergone a kidney transplant procedure.
* End-stage chronic kidney failure.
* History of heart valve abnormalities.
* Congenital heart disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-07-24 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
pNGAL concentration | 2 days
  pNGAL measurement using ELISA at baseline (before intervention) and 48 hr after intervention

SECONDARY OUTCOMES:
Mechanical Ventilation Duration | from the first day mechanical ventilation usage until weaned to T-piece, assessed up to 28 days
  Measuring hours usage of mechanical ventilation
Length of stay in ICU | 28 days
  length of stay in days during and after deresuscitation until the patient meets the ICU discharge criteria
Renal Replacement Therapy | 28 days
  Necessity of renal replacement therapy within 28 days in ICU: needed/ not
Fluid Balance (Daily) | 28 days
  Data extracted from medical record
Lactate Concentration | 2 days
  Lactate measurement from blood sample at baseline level (before intervention) and 48 hours after deresuscitation
Central Venous Pressure | 2 days
  Central venous pressure measurement using central vein catheter every 6 hours during deresuscitation
28 days mortality | 28 days
  mortality within 28 days admission to ICU: deceased or survived
Total Body Water (TBW) | 2 days
  Total Body Water measured using Bioelectrical Impedance Analysis. The total body water consists of Extracellular Water (ECW) and Intracellular Water (ICW). Measurements are conducted at baseline (before intervention) and 48 hr after intervention.
Extracellular Water (ECW) | 2 days
  Extracellular Water (ECW) using Bioelectrical Impedance Analysis. Measurements are conducted at baseline (before intervention) and 48 hr after intervention.
Intracellular Water (ICW) | 2 days
  ICW measured using Bioelectrical Impedance Analysis. Measurements are conducted at baseline (before intervention) and 48 hr after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Dita Aditianingsih, M.D, Ph.D, Principal Investigator — Indonesia University
Locations (1):
- Rumah Sakit Cipto Mangunkusumo, Jakarta Pusat, DKI Jakarta, Indonesia